CLINICAL TRIAL: NCT03407625
Title: Foley Bulb With Oral Misoprostol Versus Oral Misoprostol for Induction of Labor: A Cluster Randomized Trial
Brief Title: Foley Bulb With Oral Misoprostol for Induction of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Emily Adhikari, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 092016-026
Record Dates: First submitted 2017-12-28; First posted 2018-01-23 (Actual); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Pregnancy; Labor, Induced
Keywords: Pregnancy; Labor Induction; Cervical Ripening
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Foley bulb plus Oral Misoprostol (Experimental): Patients will received initial transcervical foley bulb, followed by oral misoprostol 100 micrograms given every 4 hours for a maximum of 2 doses.
  Interventions: Other: Foley bulb plus Oral Misoprostol
- Oral Misoprostol (Active Comparator): Patients will receive oral misoprostol 100 micrograms given every 4 hours for a maximum of 2 doses.
  Interventions: Other: Oral Misoprostol

INTERVENTIONS:
Other: Foley bulb plus Oral Misoprostol — Although labeled "experimental" for comparison purposes, this is not an experimental intervention, as the method is a currently accepted standard of care for cervical ripening and labor induction in the United States.
  Arms: Foley bulb plus Oral Misoprostol
Other: Oral Misoprostol — Patients will receive standard oral misoprostol 100mcg according to current Labor Induction Protocol.
  Arms: Oral Misoprostol

SUMMARY:
Induction of labor is associated with increased cesarean delivery rates, particularly in women with an unfavorable cervix. Both pharmacologic and mechanical methods are utilized for cervical ripening and labor induction. Evidence on the safety and effectiveness of various mechanical and pharmacologic methods of cervical ripening and labor induction is abundant, and yet the majority of clinical trials evaluate time to delivery, rather than mode of delivery. This is a prospective, cluster-randomized clinical trial to compare a standard method of induction at our institution (oral misoprostol) with an alternative, commonly used combination method of oral misoprostol and transcervical foley bulb in women with term pregnancies requiring induction of labor.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the use of a transcervical foley catheter, in combination with the standard oral misoprostol regimen will result in a decreased primary cesarean delivery rate among women with a cervical dilation of 2 centimeters of less who require induction of labor at term. This study is not an FDA-regulated study: there is no intent to test the foley bulb under an FDA-regulated protocol. Likewise, there is no intent to submit the results of this study for a change in the labeling of the foley used for this study. This study was approved by the Institutional Review Board of the University of Texas Southwestern Medical Center, and by the Office of Research Administration at Parkland Health and Hospital System.

This will be a prospective, cluster-randomized trial comparing two accepted methods of induction of labor at term among women who present for delivery at Parkland Hospital. Eligible participants will include nulliparous and multiparous women at 37 weeks gestation or greater, with a living, singleton fetus and no major fetal malformations, in cephalic presentation, with intact membranes, no prior uterine scar, who qualify for prostaglandin administration and who have a cervical dilation of 2 centimeters or less, measured at the level of the internal os. Patients with latex allergy, non-reassuring fetal status, HIV, active herpes outbreak, a prior uterine scar, or any contraindication to prostaglandins (including 4 or more painful contractions per 10 minutes prior to prostaglandin administration) will be excluded from participation in the study.

Computer-generated cluster randomization will occur on a weekly basis for all study participants, to either the combination method of foley bulb plus oral misoprostol regimen (study group) or to oral misoprostol alone regimen (control).

According to the randomization protocol each week, participants will be randomized to either the standard of care (oral misoprostol/control group) or standard of care plus foley bulb (study group). The study group will undergo placement of a 30 French foley catheter filled with 30-35cc sterile saline into the cervix in addition to the standard regimen of oral misoprostol 100 micrograms given every 4 hours for a maximum of 2 doses, for patients who meet criteria for fetal well-being, and do not had more than 4 painful contractions in 10 minutes. Misoprostol will not be administered to patients who have progressed to active labor, defined as 4 centimeters cervical dilation. The control group will undergo induction with our current standard oral misoprostol protocol alone, administered as 100 micrograms given every 4 hours for a maximum of 2 doses. Both groups will receive oxytocin as indicated by current labor protocols at our institution.

The primary outcome will be the rate of vaginal delivery. Secondary outcomes will include obstetric outcomes, maternal outcomes, and neonatal outcomes. Obstetric outcomes will include indication for induction, need for oxytocin, indication for cesarean delivery, time to active labor, time to delivery, labor analgesia, presence of chorioamnionitis, meconium-stained amniotic fluid, terbutaline use, tachysystole (defined as 6 or more contractions in 10 minutes or tetanic contraction of 120 seconds or longer) or hyperstimulation syndrome (defined as tachysystole accompanied by fetal heart rate decelerations). Maternal outcomes will include estimated blood loss, transfusion requirement, postpartum fever, uterine rupture, and unplanned hysterectomy. Neonatal outcomes will include umbilical cord blood pH, 5-minute APGAR score, intubation or ventilation in the delivery room, neonatal sepsis, and admission to Neonatal Intensive Care Unit (NICU) admission.

ELIGIBILITY:
Inclusion Criteria:

* 37 weeks gestation or greater
* Living, singleton fetus
* No major fetal malformations
* Cephalic presentation
* No prior uterine scar
* Intact fetal membranes
* Qualifies for prostaglandin administration according to current Parkland protocol
* Have a cervical dilation of 2 centimeters or less, measured at the level of the internal os
* Have an indication for induction or attempted induction of labor according to Parkland protocol

Exclusion Criteria:

* latex allergy
* non-reassuring fetal status
* HIV
* active herpes outbreak
* Prior uterine scar
* Contraindication to prostaglandins according to current Parkland protocol
* Contraindication to vaginal delivery

Min Age: 10 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2227 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily H Adhikari, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health and Hospital Systems, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adhikari EH, Nelson DB, McIntire DD, Leveno KJ. Foley Bulb Added to an Oral Misoprostol Induction Protocol: A Cluster Randomized Trial. Obstet Gynecol. 2020 Nov;136(5):953-961. doi: 10.1097/AOG.0000000000004123. PMID 33030881

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Started | 1117 | 1110
Completed | 1117 | 1110
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol | Total
Number analyzed (Participants) | 1117 | 1110 | 2227
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (6.6) | 26.6 (6.7) | 26.7 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1117 | 1110 | 2227
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black, non-Hispanic | 192 | 186 | 378
  White, non-Hispanic | 41 | 40 | 81
  Hispanic | 840 | 860 | 1700
  Other | 44 | 24 | 68
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1117 | 1110 | 2227
Parity [Count of Participants; unit: Participants]
  Parity = 0 | 591 | 584 | 1175
  Parity = 1 | 219 | 208 | 427
  Parity = 2 | 158 | 155 | 313
  Parity = > 2 | 149 | 163 | 312
Body mass index (kg/m2) [Mean (Standard Deviation); unit: kg/m^2] | 29.7 (6.7) | 30.1 (7.2) | 29.9 (7.0)
Diabetes [Count of Participants; unit: Participants]
  None | 977 | 952 | 1929
  Gestational | 99 | 115 | 214
  Pregestational | 41 | 43 | 84
Gestational age at delivery (weeks) [Median (Inter-Quartile Range); unit: weeks] | 39 [38 to 40] | 39 [38 to 40] | 39 [38 to 40]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Vaginal Delivery
Description: vaginal delivery at first induction
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1,117 | 1,110
Participants | 869 | 860
Statistical Analysis 1: Comparison: Foley Bulb Plus Oral Misoprostol vs Oral Misoprostol; Test type: Superiority; p = 0.86, log binomial regression; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.95 to 1.05]; We used generalized estimating equations for the log binomial regression with cluster entered as a random effect

2. Secondary Outcome: Time to Delivery
Description: Time (in hours) from start of induction agent to delivery at first induction
Time Frame: from start of induction agent to time of delivery
Population: This number represents women delivered at first induction
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1088 | 1075
hours | 17.3 (9.2) | 18.2 (9.2)

3. Secondary Outcome: Indication for Cesarean Delivery
Description: Among women delivered by cesarean, the indication for cesarean
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1117 | 1110
Participants
  Labor dystocia | 122 | 110
  Abnormal fetal heart rate tracing | 110 | 115
  Malpresentation | 3 | 3
  No cesarean delivery | 882 | 882

4. Secondary Outcome: Dose of Oxytocin Given (mcg or mg)
Description: Total dose of oxytocin given for induction as calculated by volume infused, concentration of solution and rate of infusion
Time Frame: at delivery
Population: Total dose of oxytocin was not found to be meaningful, thus data were not collected.
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time With Foley Bulb in Place
Description: time (in hours) from insertion to removal or expulsion of foley bulb
Time Frame: From time of documented insertion until the time of documented expulsion or removal, whichever came first, assessed up to 24 hours.
Population: Number of women with successful Foley bulb placement
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 945 | 0
hours | 5.3 [4.6 to 8.3] |

6. Secondary Outcome: Presence of Chorioamnionitis
Description: Intrapartum fever (temp equal or greater than 38C) with no other identified cause
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1117 | 1110
Participants | 203 | 155

7. Secondary Outcome: Use of Intravenous Analgesia During Labor
Description: Intravenous analgesia used between the start of induction and delivery
Time Frame: at delivery
Population: Intravenous analgesia was not clinically meaningful and was not collected
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants Used Neuraxial Analgesia During Labor
Description: Regional or neuraxial analgesia (labor epidural or spinal) used between the start of induction and delivery
Time Frame: from start of induction to delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1117 | 1110
Participants | 949 | 935

9. Secondary Outcome: Number of Participants Used General Anesthesia for Delivery
Description: General anesthesia administered for delivery
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1117 | 1110
Participants | 29 | 24

10. Secondary Outcome: Number of Participants With Meconium-stained Amniotic Fluid
Description: Identification of any meconium (green tinge) in the amniotic fluid before or during delivery by a healthcare provider's assessment of gross fluid color.
Time Frame: At the time of rupture of membranes and at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1117 | 1110
Participants | 227 | 234

11. Secondary Outcome: Terbutaline Use
Description: Administration of terbutaline, a tocolytic agent, for tetanic contractions with or without fetal heart rate decelerations
Time Frame: at delivery
Population: Terbutaline use was not felt to be clinically meaningful, and thus data were not collected
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Participants With Tachysystole
Description: 6 or more contractions in 10 minutes or tetanic contraction of 120 seconds or longer
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1117 | 1110
Participants | 325 | 313

13. Secondary Outcome: Number of Participants With Uterine Hyperstimulation Syndrome
Description: Tachysystole accompanied by fetal heart rate decelerations
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1117 | 1110
Participants | 184 | 147

14. Secondary Outcome: Number of Participants With Excess Blood Loss
Description: Maternal excess blood loss is defined as >500ml for vaginal and >1000ml for cesarean delivery
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1117 | 1110
Participants | 215 | 223

15. Secondary Outcome: Number of Participants With Blood Transfusion
Description: administration of blood products related to delivery blood loss
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1117 | 1110
Participants | 37 | 33

16. Secondary Outcome: Number of Participants With Uterine Rupture
Description: spontaneous separation of myometrium in a previously intact, unscarred uterus
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1117 | 1110
Participants | 0 | 1

17. Secondary Outcome: Number of Participants With Unplanned Hysterectomy
Description: unplanned removal of the uterus following delivery of the fetus
Time Frame: at discharge from the hospital following delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1117 | 1110
Participants | 1 | 0

18. Secondary Outcome: Number of Participants With Postpartum Fever
Description: Fever recorded in the time after delivery but prior to discharge from the hospital, with clinical assessment of endometritis
Time Frame: Following delivery and prior to discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1117 | 1110
Participants | 11 | 3

19. Secondary Outcome: Number of Participants With Umbilical Cord Blood pH <7.0
Description: Arterial or venous cord blood pH defined as <7.0
Time Frame: at delivery
Population: This number represents available umbilical cord blood gas
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1085 | 1088
Participants | 3 | 4

20. Secondary Outcome: Number of Participants With an 5-minute Apgar Score Less Than 4
Description: Appearance, Pulse, Grimace, Activity, Respirations - scored from 0 to 2 for each component, added to make a total score and used as an assessment of initial response to newborn resuscitation, lower scores associated with poor outcomes. Here defined as Apgar less than 4 at 5 minutes.
Time Frame: 5 minutes after time of birth
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1117 | 1110
Participants | 4 | 4

21. Secondary Outcome: Number of Participants That Needed Mechanical Ventilation in Delivery Room (Yes/No)
Description: Intubation with mechanical support or control of neonatal breathing in delivery room
Time Frame: at delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1117 | 1110
Participants | 2 | 4

22. Secondary Outcome: Number of Participants Administered Neonatal Antibiotics and/or Neonatal Blood Cultures
Description: Administration of neonatal antibiotics and/or neonatal blood cultures
Time Frame: From time of birth until the time of discharge or up to 7 days of life, whichever comes first.
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1117 | 1110
Participants | 277 | 237

23. Secondary Outcome: Number of Participants With Neonatal Sepsis
Description: Neonatal bacteremia as defined by bacterial growth in blood cultures
Time Frame: From time of birth until the time of discharge or up to 7 days of life, whichever comes first.
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1117 | 1110
Participants | 2 | 1

24. Secondary Outcome: Number of Participants With NICU Admission Order
Description: Admission order to neonatal intensive care unit (NICU) placed between the time of delivery and infant discharge
Time Frame: From time of birth until the time of discharge or up to 7 days of life, whichever comes first.
Measure: Count of Participants; unit: Participants
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
Number analyzed (Participants) | 1117 | 1110
Participants | 16 | 17

ADVERSE EVENTS:
Time Frame: From delivery to hospital discharge
Description: The risk of transcervical foley bulb is minimal, and the primary risk of participation in the study is breach of confidentiality. Risk associated with Foley bulb is not increased above the risks associated with vaginal or cesarean delivery; adverse maternal and neonatal outcomes are reported as secondary outcomes in this study.
Arm/Group | Foley Bulb Plus Oral Misoprostol | Oral Misoprostol
All-Cause Mortality (participants affected / at risk) | 0/1117 | 0/1110
Serious Adverse Events (participants affected / at risk) | 0/1117 | 0/1110
Other Adverse Events (participants affected / at risk) | 0/1117 | 0/1110

LIMITATIONS AND CAVEATS:
Pre-specified outcomes (dose of Oxytocin give at the delivery, terbutaline use, and the number of participants with intravenous analgesia during labor) were not collected as they were found to be not meaningful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT03407625/Prot_SAP_000.pdf